CLINICAL TRIAL: NCT07339696
Title: DANISH TITLE: Projekt Rette hjælp Til børn Med ADHD Eller Udfordringer Med Uro og Koncentration
Brief Title: Danish Access to Support and Help (DASH): Increasing Access to an Evidence-based Intervention for Children With ADHD and Their Parents
Acronym: DASH
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 152531; 152531 (Other Grant/Funding Number: TrygFonden, Denmark)
Record Dates: First submitted 2025-11-14; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: ADHD - Attention Deficit Disorder With Hyperactivity; Attention Concentration Difficulty
Keywords: ADHD parent training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NFPP-CIM Implementation Group: The group includes families with children aged 3-12 years with ADHD or attention and activity difficulties, as well as community practitioners, managers, and other local stakeholders involved in delivering the New Forest Parenting Programme - Community Implementation Model (NFPP-CIM). The study evaluates the feasibility, acceptability, and perceived outcomes of implementing NFPP-CIM in municipal child and family services.
  Interventions: Behavioral: New Forest Parenting Programme

INTERVENTIONS:
Behavioral: New Forest Parenting Programme — Parent training for children who has difficulties with attention and activity or ADHD

SUMMARY:
The aim of this study is to devise implementation strategies for the New Forest Parenting Programme (NFPP) to support a community implementation model (NFPP-CIM) and test its feasibility and acceptability for parents and stakeholders.

DETAILED DESCRIPTION:
Background Attention-deficit/hyperactivity disorder (ADHD) is a common neurodevelopmental condition associated with substantial individual and societal costs. Although effective behavioural interventions such as the New Forest Parenting Programme (NFPP) are available, access to evidence-based parent training remains limited in community settings. The current study addresses the gap between research and practice by supporting the implementation of NFPP within local Child and Family Services in Danish municipalities.

Purpose and Rationale The primary aim of this study is to develop and evaluate the feasibility and acceptability of a community implementation model for the New Forest Parenting Programme (NFPP-CIM). The project is designed as a Hybrid Type II feasibility study, focusing on both implementation processes and perceived effects in real-world community contexts. The study seeks to determine whether the NFPP-CIM can support feasible, acceptable, and sustainable delivery of NFPP by local practitioners, thereby informing future large-scale implementation.

Objectives

The study objectives are guided by the Expert Recommendations for Implementing Change (ERIC) framework and include:

To develop an NFPP Community Implementation Model (NFPP-CIM) tailored to Danish municipal contexts.

To assess the feasibility and acceptability of the NFPP-CIM among families of children with ADHD or difficulties related to attention and activity regulation, as well as among community-level stakeholders (e.g. practitioners and managers).

To explore perceived changes in family functioning and everyday life associated with participation in NFPP-CIM, and to consider how these experiences align with findings previously reported in specialist settings.

Study Design and Setting The study will employ a pre-post hybrid effectiveness-implementation design. NFPP-CIM will be delivered in three Danish municipalities by trained community practitioners in collaboration with local child and family services. Quantitative and qualitative data will be collected to examine implementation outcomes and user experiences. The project emphasizes co-creation, user participation, and interagency collaboration to strengthen local ownership and sustainability.

Implementation Outcomes Consistent with the study's implementation focus, feasibility and acceptability constitute central outcomes of the project.

Feasibility of implementing the NFPP-CIM will be assessed using quantitative implementation indicators, including:

Recruitment rate, defined as the proportion of eligible families who consent to participate (assessed from initial contact to enrollment).

Completion rate, defined as the proportion of enrolled families who complete the intervention and post-intervention assessment.

Practitioner adherence, defined as fidelity to the NFPP-CIM manual, assessed through session checklists completed throughout the intervention period (approximately 16 weeks).

Acceptability of the NFPP-CIM will be examined using qualitative methods, including semi-structured interviews and brief open-ended satisfaction questionnaires completed by parents. These data will explore the perceived practicality, usefulness, and overall experience of participating in the intervention. Acceptability data will be collected at post-intervention, within six weeks after completion of the programme.

Expected Outcomes and Significance Findings will provide insight into how NFPP can be effectively implemented and scaled up in community settings. Specifically, the study will inform refinement of NFPP training models for local practitioners, strategies for user involvement, and approaches to sustaining cross-sector collaboration. By focusing on real-world feasibility and stakeholder experiences, the study aims to bridge the gap between evidence-based ADHD interventions and community-based practice and to support improved access to high-quality services for families.

ELIGIBILITY:
Inclusion Criteria:

* Families receiving services through municipal child and family clinics in Denmark
* Child aged 3-12 years
* Parent-perceived difficulties with attention and activity regulation, including those with a diagnosis or suspected diagnosis of ADHD.
* All custodial parents willing and able to provide informed consent
* Parents interested in participating in the New Forest Parenting Programme - Community Implementation Model (NFPP-CIM)

Exclusion Criteria:

* Families not receiving services through municipal child and family clinics
* Parents unable to provide informed consent
* Families unable to participate in the intervention due to severe child or family circumstances that preclude engagement (e.g. acute crisis requiring alternative services, Parents or children with severe mental or physical illness that would prevent active participation in the intervention)

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population includes families receiving services through municipal child and family clinics in Denmark. Participating families have children aged 3-12 years who present with parent-perceived difficulties related to attention and activity regulation, including diagnosed or suspected ADHD. All custodial parents provide informed consent and complete the quantitative outcome measures.
  In addition, the study includes community practitioners, managers, and other stakeholders involved in delivering and supporting the New Forest Parenting Programme - Community Implementation Model (NFPP-CIM). These participants complete semistructured interviews and contribute qualitative data related to feasibility, acceptability, and implementation processes and do not complete quantitative outcome questionnaires (see detailed study description).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome (exploratory clinical signal): ADHD Rating Scale-IV (ADHD-RS-IV) Danish Version - parent ratings | Change in ADHD symptoms measured by ADHD-RS from baseline to post-intervention. I.e. From T1: enrolment (baseline) to T2: T2 (End of treatment): approximately 16 weeks after T1 to T3 (Follow-up): approximately 36 weeks after T2.
  This outcome is included solely as an exploratory signal of change to inform the design of a future fully powered trial; the current study is not powered to detect statistically significant effects.The ADHD-RS is an 18-item questionnaire that addresses child symptoms of ADHD and symptoms of oppositional defiant disorder/conduct disorder on a four point scale ('not at all' to 'very often') (DuPaul, G.J., et al., Parent ratings of attention-deficit/hyperactivity disorder symptoms: Factor structure and normative data. Journal of Psychopathology and Behavioral Assessment, 1998. 20(1): p. 83-102.)

SECONDARY OUTCOMES:
The Strengths and Difficulties Questionnaire (SDQ) - Danish parent version | Change in SDQ scores from baseline (T1) at enrollment, to post-intervention (T2) approximately 16 weeks after T1, and to follow-up (T3) approximately 36 weeks after T2.
  The Strengths and Difficulties Questionnaire (SDQ) is a brief, validated screening measure of emotional and behavioural difficulties in children and adolescents aged 2-17 years. It consists of 25 items rated on a 3-point scale (0 = Not true, 1 = Somewhat true, 2 = Certainly true). The following scores are used in this study:
  - Total Difficulties Score: Sum of four subscales (Emotional Symptoms, Conduct Problems, Hyperactivity/Inattention, Peer Problems; 20 items).
  Score range: 0-40. Higher scores indicate greater difficulties (worse outcome).
  * Conduct Problems Subscale: Five items assessing behavioural difficulties. Score range: 0-10. Higher scores indicate greater conduct problems (worse outcome).
  * Impact Score (SDQ Impact Supplement): Assesses perceived distress and functional impairment related to the child's difficulties in everyday life.
  Score range: 0-10. Higher scores indicate greater impact and impairment (worse outcome).
The Parenting Sense of Competence Scale (PSOC) Danish version - parent ratings | Change in PSOC scores from baseline (T1) at enrollment, to post-intervention (T2) approximately 16 weeks after T1, and to follow-up (T3) approximately 36 weeks after T2.
  The Parent Sense of Competence Scale (PSOC) is a widely used questionnaire assessing parents' perceived competence in their parenting role. There are separate mother and father versions of the PSOC. The PSOC consists of 16 items rated on a 6-point Likert scale (from strongly disagree to strongly agree) and yields two subscale scores:
  Satisfaction subscale: 9 items assessing parental satisfaction, anxiety, motivation, and frustration.
  Efficacy subscale: 7 items assessing perceived parenting competence, capability, and problem-solving ability.
  Score range:
  Total score: 16-96 (Satisfaction and Efficacy subscales scored separately)
  Interpretation:
  Higher scores indicate greater parental competence and confidence / better outcome.
Family Strain Index (FSI) - parent ratings | Change in FSI scores from baseline (T1) at enrollment, to post-intervention (T2) approximately 16 weeks after T1, and to follow-up (T3) approximately 36 weeks after T2.
  The Family Strain Index (FSI) is a 6-item questionnaire measuring the impact of the child's ADHD-related difficulties on family life, including stress, strain, and burden.
  Score range: 0-24 Interpretation: Higher scores indicate greater family strain and burden / worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette Lange, Principal Investigator — Aarhus University Hospital
Locations (1):
- Forskningsafdelingen - Børne- og Ungdomspsykiatrisk Afdeling, Psykiatrien-Skejby, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to data protection regulations

REFERENCES:
- [Background] Alexandre, J.L., et al., The ADHD rating scale-IV preschool version: Factor structure, reliability, validity, and standardisation in a Danish community sample. Research in Developmental Disabilities, 2018. 78: p. 125-135. Arnfred, J., et al., Danish norms for the Strengths and Difficulties Questionnaire. Danish medical journal, 2019. 66(6). Borrelli, B., The assessment, monitoring, and enhancement of treatment fidelity in public health clinical trials. 2011. p. S52-S63. Bowen, D.J., et al., How we design feasibility studies. American journal of preventive medicine, 2009. 36(5): p. 452-457. Cohen, A.N., et al., Improving care quality through hybrid implementation/effectiveness studies: Best practices in design, methods, and measures. Implementation Science, 2015. 10(1): p. A29. Curran, G.M., et al., Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Medical care, 2012. 50(3): p. 217. Damschroder, L.J., et al., Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implementation Science, 2009. 4(1): p. DuPaul, G.J., et al., Parent ratings of attention-deficit/hyperFactor structure and normative data. Journal of Psychopathology and Behavioral Assessment, 1998. 20(1): p. 83-102. Fixsen, D., et al., Statewide implementation of evidence-based programs. Exceptional children, 2013. 79(2): p. 213. Fixsen, D., et al., Statewide implementation of evidence-based programs. Exceptional Children, 2013. Goodman, R., et al., Using the Strengths and Difficulties Questionnaire (SDQ) to screen for child psychiatric disorders in a community sample. The British Journal of Psychiatry, 2000. 177(6): p. 534.